CLINICAL TRIAL: NCT04791449
Title: Exercise Enhances Wound Healing in Patients With Diabetic Foot Ulcers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Responsible Party: Principal Investigator, Eric J Lew, Dr. Eric J. Lew, MD, University of New Mexico
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19-537
Record Dates: First submitted 2021-03-04; First posted 2021-03-10 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Intervention Model Description: This study is based on a two-group repeated measures design.
Who Masked: Care Provider
Masking Description: Podiatrist and wound care technician will be blinded to an individual's participation and group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment-as-usual plus medically-supervised exercise (TAU-EX) (Experimental): This group attends normal wound care appointments as scheduled with the wound care provider, generally 2 - 3 times per week. Coincident with these appointments, ideally, they will also attend a medically-supervised exercise program supervised by the exercise physiologists of the Cardiac Rehabilitation facility. The exercise sessions will last no more than 1-hr per session. The maximum number of sessions possibly attended over the 12-wk intervention period is 36. In addition, participants in this group will maintain their activities of daily life unless contraindicated by the would care provider.
  Interventions: Other: Structured exercise program
- Treat-as-usual (TAU) (No Intervention): This group attends normal wound care appointments as scheduled with the wound care provider, generally 2 - 3 times per week. In addition, participants in this group will maintain their activities of daily life unless contraindicated by the would care provider.

INTERVENTIONS:
Other: Structured exercise program — Medically-supervised participation in 2-3 exercise sessions per week over 12-wk study period. Exercise conducted in the cardiac rehabilitation program.
  Arms: Treatment-as-usual plus medically-supervised exercise (TAU-EX)

SUMMARY:
The overarching purpose of this study is to investigate the impact that exercise, as delivered through a medically supervised, outpatient cardiac rehabilitation program, has on the wound healing process in Type 2 diabetics having foot ulcers classified as being Wound, Ischemia, foot Infection (WIfI) stage 2 or lower. The criterion reference measure of diabetic foot ulcer wound healing is be the time required to reach the maturation phase of the wound healing cascade (wound closure without drainage).

DETAILED DESCRIPTION:
This study uses a two-group repeated measures design. Sixty volunteers will be recruited through the University of New Mexico (UNM) Center for Healing in the Lower Extremity (CHILE) clinic. A letter explaining the study will be placed in the file of all diabetic foot ulcer (DFU) clients of CHILE clinic. There is section to be completed by interested clientele (RSVP) and placed it in labelled box in the clinic office.

A research team member collects box contents (M-F) and contacts all respondents using the preferred method provided on the RSVP to conduct an initial screening of inclusion/exclusion criteria and review study requirements. Those not qualifying for the study or uninterested will be thanked for their initial interest. If the respondent is a viable prospect for inclusion, the electronic medical record will be reviewed by the authorized research team member to verify inclusion criteria are satisfied and no exclusion criteria are present. An initial study-related appointment coinciding with their next scheduled wound care appointment at the CHILE clinic will be set for eligible prospects. After screening into the study, the prospects will be randomly assigned to a group via an online randomizer. Group 1 (Treatment as Usual, TAU) participants receive the regularly scheduled standard wound care. Group 2 (Treatment as Usual plus Exercise, TAU-EX) receives the regularly scheduled standard wound care and is assigned to the 12 -week medically supervised exercise program. Body mass index (BMI), HbA1c, weight (wearing similar clothes at each weigh in), and vascular endothelial growth factor (VEGF) levels will be measured at baseline and then again at 4, 8 and 12 weeks.

The Informed Consent will be provided for the prospect's review; questions asked of the research team member are encouraged. The 50:50 likelihood of being randomly assigned to one of two groups (TAU or TAU-EX) will be explained. All participants will receive their regularly scheduled standard wound care (per CHILE Clinic procedures) 2-3 times a week for 12 weeks or until the wound healed if less than 12 weeks. Expectations of group assignment and incentivizing prospects for their time will be discussed fully. If the prospect wants to continue with the study, the Informed Consent will be signed. If the prospect does not want to continue, they will be thanked for their time plus encouraged to continue with their scheduled wound care appointments and follow their wound care professional's recommendations. A Spanish interpreter, in person or via phone, will be used for all subjects who are not fluent in English. Official Spanish language versions of the Consent Form and study questionnaires will be available as well. Regardless of group assignment, the participant will be reminded to continue with their normally scheduled wound care appointments and to follow their wound care professional's recommendations. All participants will also be encouraged to maintain their normal daily activities unless contraindicated by their wound care provider. A typical wound care appointment consists of the CHILE clinic wound care technician removing the dressing. A wound care provider evaluates the drainage and the wound. It is then cleaned with Vashe (Steadme Medical, Fort Worth, TX). The periwound is cleaned with Hibiclens (Molnlycke Health Care, Brooklyn, NY). If debridement is necessary, it is performed by the wound care provider as appropriate for the tissue type and location. Measurement of the wound will be done weekly by the wound care provider using one of two accepted wound measurement methods - clock method or modified clock method. Deviations from the 12:00 - 6:00 numbering scheme are documented for length (i.e 2:00 - 8:00) and width at the widest perpendicular (i.e. 10:00 - 5:00) point to the line of length. Wound depth will be measured at the deepest section and any undermining or tunneling will be referred to by the clock measures. New dressings will be applied.

After giving written consent, the TAU-EX participant will be scheduled for an initial intake session at the UNM Cardiac Rehabilitation facility (ground floor of UNM hospital, UNMH) to review risk factors, current exercise habits, exercise session expectations and undergo a program orientation. They will sign a second consent form, be given a tour of the facility and familiarized with the exercise equipment. They will be reminded that they will be exercising along with cardiac rehabilitation clients in 2 to 3 exercise sessions per week; the sessions will ideally coincide with the TAU-EX participant's normally scheduled wound care appointments. An appointment will be scheduled so the Cardiac Rehabilitation staff can conduct a maximal exercise capacity test per the facility's standard procedure (note: arm-ergometry will be used); the heart rate (HR), blood pressure (BP), rating of perceived exertion (RPE), arm cranking cadence and intensity will be converted to MET (metabolic equivalent of task) level(s) with peak MET (MET peak) being the basis for each individualized exercise prescription. Systematic program progression is supervised by the cardiac rehabilitation program staff. Exercise program adjustments to intensity, duration, and modality will be made each session as appropriate and as tolerated by the participant. Exercise-related variables (i.e. intensity, duration, and modality) will be recorded each session. HR and oxygen saturation (O2 sat) will be recorded pre-, during and post exercise. Blood pressure and non-fasting blood glucose will be recorded pre- and post-exercise.

The first exercise session begins with a pre-participation non-fasting blood glucose finger stick, resting HR and BP assessments, a brief (e.g. 5-minute) warm-up on an arm ergometer, and a consult regarding session goals. The exercise physiologist will encourage the participant to exercise in timed bouts at the combination of cadence and resistance equivalent to 50% of MET peak. Each bout is followed by a recovery period (low speed cadence, very light resistance) until HR approaches the pre-exercise level. This is followed by iterations of exertion and active recovery until 20-30 minutes have passed. Following the last bout's active recovery period and seated rest for hemodynamic assessment, the exercise physiologist records all session data, comments, observations, and reviews the session with the participant before scheduling the next exercise session. All subsequent exercise sessions begin with a pre-participation finger stick (blood glucose target range is 100-250 mg/dL), resting hemodynamic assessment, brief warm-up, and consult. Together the exercise physiologist and participant set new goals for the day's session (i.e. increase cadence by 10 rpm at same resistance, exercise at the RPE associated with a slightly higher intensity, add 20 seconds to the exercise bout for the session, etc.). The participant's physiological responses are monitored to ensure safety and recorded for use in upcoming sessions. Exercise prescriptions will be progressed based on individual tolerance, adaptation, and motivation.

Standard wound care appointments consist of removal of wound dressing, evaluation of wound (e.g. drainage, tissue status), wound cleaning, debridement as necessary, measurement, redressing, and offloading (e.g. total contact casting), as applicable. Over the 12-wk intervention period, all participants will be instructed to continue their normal daily routines and adherence to the podiatrist's recommendations. The blood glucose range of 100-250 mg/dL is the acceptable range for the participant to be able to begin the day's exercise program. If the glucose is above or below that range and the participant is symptomatic, the clinic staff will contact the designated research team member who will contact the participant's primary care provider and either refer them to their services or direct the staff to take them to the UNM Urgent Care Clinic. If the participant is asymptomic, the clinic staff will contact the designated research team member and she will discuss the options with the participant regarding going home and re-adjusting meals, medication, or whatever seemed to be the problem and have the participant return to exercise in 1-2 days.

Volunteers may withhold participation or withdraw from the study at any time without impact on their DFU wound care at the CHILE clinic; coverage of TAU-EX exercise sessions will cease. Participants may be withdrawn from the study by research team members if instructions are repeatedly ignored or the participant is deemed at risk for harming themselves if they continue. Upon withdrawal from the study, any hard copy information will be placed in a locked medical records bin that is destroyed in accordance with UNM hospital regulations for destroying all patient information. Data collected prior to withdrawal will remain in the study database and may not be removed until 6 years after the study is completed.

As with any type of exercise, there are risks of injury, loss of consciousness, heart attack and death. Unaccustomed increases in HR, breathing rate, and sweating during exercise sessions, self-consciousness when exercising in a small group, and muscle soreness are all normal responses to exercise. Development of an infection may or may not be associated with the exercise program. All in the TAU-EX group will have provided documentation indicating their medical provider approved of their participation. TAU-EX members will be counseled regarding the warning signs and symptoms of heart attacks, shortness of breath, and/or loss of consciousness.

All exercise sessions will be supervised by the exercise physiologists of the UNMH cardiac rehabilitation program; symptoms indicative of cardiometabolic distress will result in stoppage or intensity reduction of the exercise session. Participants in the TAU and TAU-EX groups may experience bruising, soreness, bleeding, fainting as a result of blood draws and discomfort resulting from the wound care appointments. Finger sticks for the TAU-EX group may result in localized discomfort and/or bruising. DFU wound care is part of each participant's normal treatment plan and beyond the scope of this study.

There may be no direct benefit for individuals participating in this study. However, some people have experienced weight loss, improved blood glucose control, and faster wound healing when exercising on a regular basis. On a larger scale, results from this study may inform the treatment plan of individuals receiving medical care for DFUs.

Based on the nature of the research and the data that will collected, The investigators may find that adherence to the wound care appointment schedules are increased for those in the TAU-EX group compared to TAU. The investigators may also find that adherence may be predicted based on some of the response combinations recorded on the questionnaires (i.e. support of partner, transportation, comradery developed during exercise sessions).

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of type 2 diabetes
* 20 - 80 years of age
* Ankle-Brachial Index (ABI) > 0.6 or Toe Pressure (TcPO2) > 40 mmHg
* recent (within 12 weeks) blood glucose value between 100 - 350 mg/dL
* recent (within 12 weeks) HbA1c value < 14 %,
* DFU of WIfI Grade 2 or less
* fluency in reading and speaking English or Spanish.

Exclusion Criteria:

* inability to provide own consent
* inability to obtain permission to participate from a medical professional
* lack of consistent mode of transportation to UNMH
* infection to any part of the body
* patients that has had a transplant and/or is immunocompromised
* prisoners.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-10-10 (Actual); Primary Completion 2035-05-31 (Estimated); Study Completion 2035-05-31 (Estimated)

PRIMARY OUTCOMES:
wound healing time | 12 weeks or less
  number of days from enrollment required to reach the maturation phase of the wound healing cascade (wound closure without drainage)

CONTACTS AND LOCATIONS:
Overall Officials: Eric J Lew, DPM, Principal Investigator — University of New Mexico Health Sciences Center
Locations (1):
- UNM Cardiac Rehabilitation Services, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bloor CM. Angiogenesis during exercise and training. Angiogenesis. 2005;8(3):263-71. doi: 10.1007/s10456-005-9013-x. Epub 2005 Nov 19. PMID 16328159
- [Background] Byrne AM, Bouchier-Hayes DJ, Harmey JH. Angiogenic and cell survival functions of vascular endothelial growth factor (VEGF). J Cell Mol Med. 2005 Oct-Dec;9(4):777-94. doi: 10.1111/j.1582-4934.2005.tb00379.x. PMID 16364190
- [Background] Colwell AS, Beanes SR, Soo C, Dang C, Ting K, Longaker MT, Atkinson JB, Lorenz HP. Increased angiogenesis and expression of vascular endothelial growth factor during scarless repair. Plast Reconstr Surg. 2005 Jan;115(1):204-12. PMID 15622252
- [Background] Keylock T, Young H. Delayed wound healing: can exercise accelerate it? International Journal of Exercise Science 3(3): 70-78, 2010.
- [Background] Riebe D. et al. ACSM's Guidelines for Exercise Testing and Prescription 10th ed. Philadelphia (PA). Wolters Kluwer; 2018.
- [Background] Eraydin S, Avsar G. The Effect of Foot Exercises on Wound Healing in Type 2 Diabetic Patients With a Foot Ulcer: A Randomized Control Study. J Wound Ostomy Continence Nurs. 2018 Mar/Apr;45(2):123-130. doi: 10.1097/WON.0000000000000405. PMID 29521922
- [Background] Arena R, Lavie CJ, Cahalin LP, Briggs PD, Guizilini S, Daugherty J, Chan WM, Borghi-Silva A. Transforming cardiac rehabilitation into broad-based healthy lifestyle programs to combat noncommunicable disease. Expert Rev Cardiovasc Ther. 2016;14(1):23-36. doi: 10.1586/14779072.2016.1107475. Epub 2015 Oct 29. PMID 26511659
- [Background] Pence BD, DiPietro LA, Woods JA. Exercise speeds cutaneous wound healing in high-fat diet-induced obese mice. Med Sci Sports Exerc. 2012 Oct;44(10):1846-54. doi: 10.1249/MSS.0b013e31825a5971. PMID 22543735
- [Background] Matos M, Mendes R, Silva AB, Sousa N. Physical activity and exercise on diabetic foot related outcomes: A systematic review. Diabetes Res Clin Pract. 2018 May;139:81-90. doi: 10.1016/j.diabres.2018.02.020. Epub 2018 Feb 23. PMID 29477503
- [Background] Emery CF, Kiecolt-Glaser JK, Glaser R, Malarkey WB, Frid DJ. Exercise accelerates wound healing among healthy older adults: a preliminary investigation. J Gerontol A Biol Sci Med Sci. 2005 Nov;60(11):1432-6. doi: 10.1093/gerona/60.11.1432. PMID 16339330
- See also: Flahr. The Effect of Nonweight-bearing Exercise and Protocol Adherence on Diabetic Foot Ulcer Healing: A Pilot Study — https://www.o-wm.com/content/effect-nonweight-bearing-exercise-and-protocol-adherence-diabetic-foot-ulcer-healing-pilot-s